CLINICAL TRIAL: NCT05346835
Title: Intermediate-Size Population Expanded Access Program (EAP) for Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS) in Patients With Multiple Myeloma
Brief Title: Expanded Access Program (EAP) for Ciltacabtagene Autoleucel (Cilta-Cel) Out-of-Specification (OOS) in Participants With Multiple Myeloma
Status: Available | Type: Expanded Access
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108968; 68284528MMY4006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-03-21; First posted 2022-04-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Cilta-cel OOS Therapy — Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS) will be provided as a one-time administration as an intravenous infusion.
  Other Names: JNJ-68284528

SUMMARY:
The purpose of this expanded access program (EAP) is to provide ciltacabtagene autoleucel (cilta-cel) that does not meet the commercial release specifications of CARVYKTI and is not available via the local health care system in the country where the treatment is requested.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for treatment with cilta-cel per United States Prescribing Information (USPI)
* Has serious or life-threatening multiple myeloma per USPI, and where re-apheresis, re-manufacturing, or other anti-myeloma directed therapy is not considered feasible or adequate per treating physician discretion
* Favorable participant benefit/risk assessment determined by Janssen medical review
* Treating physician confirms the favorable risk benefit profile, and that proceeding with this treatment is in the best interest of the participant
* Able to provide informed consent indicating they understand the purpose of this expanded access program (EAP)
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test during screening and prior to the first dose of cyclophosphamide and fludarabine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (137):
- United States (136):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cancer Treatment Center of America Phoenix, Goodyear, Arizona
  - HonorHealth Cancer Transplant Institute, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - The University of Arkansas for Medical Sciences Myeloma Institute for Research and Therapy, Little Rock, Arkansas
  - Alta Bates Medical Center Cancer Center, Berkeley, California
  - City of Hope, Duarte, California
  - University of California at San Diego, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Center Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles UCLA, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Sutter Medical Foundation, Sacramento, California
  - University of Calif Davis Medical Center, Sacramento, California
  - UCSF, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - UCHealth Cancer Care Anschutz Medical Campus University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Care, Newark, Delaware
  - MedStar Georgetown Hospital, Washington D.C., District of Columbia
  - University of Florida at Shands, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute at Baptist Health / Baptist Health Medical Group, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Tampa General Hospital, Tampa, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - City of Hope Cancer Center, Newnan, Georgia
  - Kapi Olani Medical Center for Women and Children Hawaii Pacific, Honolulu, Hawaii
  - St. Luke's Mountain State Tumor Institute, Boise, Idaho
  - Northwestern Medicine - Northwestern Memorial Hospital Galter Pavilion, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University Of Illinois, Chicago, Illinois
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - NorthShore University Health System, Evanston Hospital, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - City of Hope Chicago, Zion, Illinois
  - IU Health University Hospital, Indianapolis, Indiana
  - St Francis Hospital & Health Centers Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Community Health Network MD Anderson Cancer Center, Kokomo, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Fairway, Kansas
  - Ascension via Christi Research, Wichita, Kansas
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University School of Medicine JHUSOM, Baltimore, Maryland
  - Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Brigham and Women's Cancer Center, Weymouth, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute - Lawrence and Idell Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - William Beaumont Health System, Royal Oak, Michigan
  - M Health Fairview University of Minnesota Medical Center East Bank, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers, The State Univ of NJ-Robert Wood Johnson Medical School-The Cancer Institute of NJ (CINJ), New Brunswick, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - The Feinstein Institute for Medical Research (Northwell Health Inc.), Manhasset, New York
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai - The Derald H. Ruttenberg, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Good Samaritan Hospital, Cincinnati, Ohio
  - The Jewish Hospital - Mercy, Cincinnati, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - James Cancer Hospital, Columbus, Ohio
  - OhioHealth Mansfield Hospital, Columbus, Ohio
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health And Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Ctr, Hershey, Pennsylvania
  - University of Pennsylvania Division of Hematology Oncology Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Avera McKennan Hospital, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Sarah Cannon Cancer Institute, Nashville, Tennessee
  - Tennessee Valley Healthcare System, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - San Antonio Methodist TX Transplant Physicians Group, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Healthcare, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Schar Cancer Institute Dept of Fairfax Hospital, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Swedish Cancer Institute First Hill, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - West Virginia University Medical Center, Morgantown, West Virginia
  - University Of Wisconsin Hospital, Madison, Wisconsin
  - Aurora Saint Lukes Medical Center, Milwaukee, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- DUMMY, Dummy, Germany